CLINICAL TRIAL: NCT00858286
Title: Follow-up Survey to Compare Stable Dosing (SERETIDE) With SYMBICORT SMART, Maintenance and Reliever Therapy in One Inhaler in Moderate and Severe Asthmatics.
Brief Title: A Follow-up Survey to Compare Stable Dosing (SERETIDE) With SYMBICORT, SMART, Maintenance and Reliever Therapy in One Inhaler in Moderate and Severe Asthmatics.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109780
Record Dates: First submitted 2009-02-19; First posted 2009-03-09 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stable dosing with SERETIDE, short acting B-2agonist as needed (Experimental): Regular treatment with SERETIDE in a stable dosing with short acting beta-2 agonists as needed
  Interventions: Other: Spirometry, PEF measurements and diary cards to evaluate control of Asthma
- Maintenance treatment with SYMBICORT and SYMBICORT as needed (Experimental): Maintenance treatment with SYMBICORT and using the same inhaler with SYMBICORT as needed
  Interventions: Other: Spirometry, PEF measurements and diary cards to evaluate control of Asthma

INTERVENTIONS:
Other: Spirometry, PEF measurements and diary cards to evaluate control of Asthma — No intervention is made with the existing therapy, but patient will perform spirometry and PEF evaluations together with a registration of control of asthma in diary cards and health economic parameters in questionnaires

SUMMARY:
The purpose with this study is to describe in detail the control or lack of control of asthma, based on two different dosing strategies, regular treatment with SERETIDE in a stable dosing with short acting beta-2 agonists as needed, or maintenance treatment with SYMBICORT and using the same inhaler with SYMBICORT as needed.

DETAILED DESCRIPTION:
The purpose with this study is to describe in detail the control or lack of control of asthma, based on two different dosing strategies. No therapy intervention is made with existing prescribed medications (SERETIDE or SYMBICORT), but evaluations outside standard care is made by evluations with diary cards, questionnaires, PEF evaluations and spirometry which is regarded as the intervention by the Swedish Authorities.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* 18 years or above
* able to fill in questionnaires and perform PEF measurements
* asthma diagnosis and prescribed SERETIDE or SYMBICORT, either regular treatment using SERETIDE in a stable dosing and short acting B2 agonists as needed, or maintenance treatment with SYMBICORT but also using same inhaler SYMBICORT as needed

Exclusion Criteria:

* no other lung disease
* neurological disease with psychological handicap
* cerebro-vascular disease with handicap
* un-stable cancer
* known or planned pregnancy during the time of the study
* subjects who have serious uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
asthma control based on GINA guidelines from 2007. | 3 months

SECONDARY OUTCOMES:
Quality of Life, Health economics and exacerbations | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Stockholm, Sweden